CLINICAL TRIAL: NCT05571787
Title: A Phase 1, Open-label, 4-period, Randomized 6-sequence Study to Evaluate the Effect of Food and Rabeprazole, a Proton Pump Inhibitor, on the Pharmacokinetics of HMPL-523 in Healthy Volunteers
Brief Title: HMPL-523 Food Effect and Proton Pump Inhibitor Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2022-523-00US1
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Relapsed or Refractory Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma | interventions — Rabeprazole

STUDY DESIGN:
Intervention Model Description: Open-label, 4-Period, Randomized 6-Sequence Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): Subjects in treatment A will fast overnight for at least 10 hours prior to HMPL-523 dosing.
  Interventions: Drug: HMPL-523
- Treatment B (Experimental): Subjects in treatment B will receive a standardized high-fat meal approximately 30 minutes before HMPL-523 administration
  Interventions: Drug: HMPL-523
- Treatment C (Experimental): Subjects in treatment C will receive a standardized low-fat meal approximately 30 minutes before HMPL-523 administration
  Interventions: Drug: HMPL-523
- Treatment D (Experimental): Subjects in treatment D will receive rabeprazol 1 hour prior to receiving a standardized low-fat meal. On Day 26 subjects will also receive HMPL-523 approximately 30 minutes after the standardized low-fat breakfast
  Interventions: Drug: HMPL-523; Drug: Rabeprazole

INTERVENTIONS:
Drug: HMPL-523 — 700 mg HMPL-523 will be administered by mouth once daily on Day 1, Day 8, Day 15, and Day 26
Drug: Rabeprazole — 40 mg of rabeprazole will be administered by mouth once daily in the morning from Day 20 to Day 26
  Arms: Treatment D

SUMMARY:
A Phase 1, Open-label, 4-Period, Randomized 6-Sequence Study to Evaluate the Effect of Food and Rabeprazole, a Proton Pump Inhibitor, on the Pharmacokinetics of HMPL-523 in Healthy Volunteers

DETAILED DESCRIPTION:
This study will be a single-center, open-label, 4-period, randomized,6-sequence study conducted with 24 healthy male or female subjects. The study will consist of a Screening Phase (Screening and Day -1), a Treatment Phase (Periods1, 2, 3,and 4), and an End of Study (EOS) Phase. Screening must occur within 28 days before the first study drug administration. There will be a washout of at least 7days between 4 administrations of HMPL-523.Subjects in Periods 1, 2, and 3 will be randomized into 1 of 6 treatment sequences, with all subjects then receiving the same treatment in Period 4.

ELIGIBILITY:
Inclusion Criteria:

1. The volunteer is male or female between the ages of 18 and 55 years old (inclusive) at the time of informed consent.
2. The volunteer has a body mass index (BMI)>18 and ≤29.9 kg/m2at screening.
3. Females must be postmenopausal (defined as absence of menses for at least 1year without alternative medical cause)or permanently sterile by total hysterectomy, bilateral oophorectomy, or bilateral salpingectomy.
4. Males, including those who have had a successful vasectomy, must use a condom during sexual intercourse with women of childbearing potential, starting from their first dose of study drug through 30 days after their last dose of study drug. Alternatively, abstinence is allowed if it is the normal and preferred lifestyle of the volunteer.
5. The volunteer must provide written informed consent prior to any study specific screening procedures.
6. The volunteer is willing and able to comply with all aspects of the protocol, as determined by the PI.

Exclusion Criteria:

1. The volunteer has a known history of any gastrointestinal surgery or any condition possibly affecting drug absorption (eg, cholecystectomy, gastrectomy, achlorhydria, peptic ulcer disease, or history of stomach or intestinal surgery or resection). Note: Appendectomy and hernia repairs are allowed.
2. The volunteer had a clinically significant illness within 8 weeks or a clinically significant infection within 4 weeks prior to the first dose.
3. The volunteer has evidence of a clinically significant deviation from normal in the physical examination, vital signs, or clinical laboratory determinations at screening or at Day -1 check-in (baseline).
4. The volunteer has systolic blood pressure >140 mmHg oradiastolic blood pressure >90mmHg.
5. The volunteer has a clinically significant ECG abnormality, including a marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTcF interval >480msec), or hasa family history of prolonged QTc syndrome or sudden death.
6. The volunteer has a history of smoking or use of nicotine-containing substances within the previous 2 months, as determined by medical history or volunteer's verbal report and confirmed by cotinine test at check-in.
7. The volunteer has a history of drug or alcohol misuse within 6 months prior to screening or a positive urine drug test at screening or at check-in.
8. The volunteer has been diagnosed with acquired immune deficiency syndrome or has performed tests that are positive for human immunodeficiency virus (HIV), HepatitisBvirus (HBV), orHepatitis C virus (HCV).
9. The volunteer has participated in a clinical trial of other study drug before screening, and the time since the last use of other study drug is less than 5 times the half-life or 4 weeks, whichever is longer, or the volunteer is currently enrolled in another clinical trial.1
10. The volunteer has consumed grapefruit, starfruit, Seville oranges, or their products within 7 days prior to the first dose.
11. The volunteer has consumed herbal preparations/medications, including, but not limited to, St. John's Wort, kava, ephedra (ma huang), Ginkgo biloba, dehydroepiandrosterone, yohimbe, saw palmetto, and ginseng, within 7 days prior to the first dose (21days for St.John's Wort).
12. The volunteer has experienced a weight loss or gain of >10% within 4 weeks prior to the first dose as noted by medical history and weight at screening and check-in.
13. The volunteer has received blood or blood products within 4 weeks, donated blood or blood products within 8 weeks prior to the first dose or donated double red cell within 16weeks prior to first dose.
14. The volunteer has used any over-the-counter (OTC) medications or prescription drugs (medications that can lower gastric acid in particular) within 2 weeks prior to the first dose.
15. The volunteer is allergic to any of the study drugs (or its excipients) to be given in this study.
16. A female participant is pregnant, lactating, or breastfeeding.
17. A male volunteer who plans to donate sperm or father a child within 30 days after receiving the study drug.
18. The volunteer has any condition that would make him or her, in the opinion of the PIor Sponsor, unsuitable for the study, or who, in the opinion of the PI, is not likely to complete the study for any reason.Note: One repeat of laboratory assessments, including vital signs and ECG,may be performed at screening and at -check-in(Day-1) at the discretion of the PI.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
PK parameter for HMPL-523: AUC0-t | Day 1 to Day 31
  Area under the concentration time curve from time 0 to the last measurable concentration
PK parameter for HMPL-523: AUC0-inf | Day 1 to Day 31
  Area under the concentration time curve from time 0 extrapolated to infinity
PK parameter for HMPL-523: Cmax | Day 1 to Day 31
  Maximum observed plasma concentration
PK parameter for HMPL-523: tmax | Day 1 to Day 31
  Time to reach the maximum observed plasma concentration

SECONDARY OUTCOMES:
Assessment of safety procedures findings | Day 1 to Day 31
  Any untoward medical occurrence associated with the study drug
PK parameter for metabolite M1: AUC0-t | Day 1 to Day 31
  Area under the concentration time curve from time 0 to the last measurable concentration
PK parameter for metabolite M1: AUC0-inf | Day 1 to Day 31
  Area under the concentration time curve from time 0 extrapolated to infinity
PK parameter for metabolite M1: Cmax | Day 1 to Day 31
  Maximum observed plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No